CLINICAL TRIAL: NCT06426706
Title: Paravertebral Block or Serratus Posterior Superior Intercostal Plane Block in Pain Management After Video-Assisted Thoracoscopic Surgery: A Randomized Controlled Clinical Trial
Brief Title: TPVB or SPSIPB in Pain Management After VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, MD, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024.174.IRB1.019
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Video-assisted Thoracoscopic Surgery; Paravertebral Block; Serratus Posterior Superior Intercostal Plane Block; Regional Anesthesia Morbidity
Keywords: video-assisted thoracoscopic surgery; paravertebral block; serratus posterior superior intercostal plane block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Participants who will be receiving a serratus posterior superior intercostal plane block with a single dose of 30 ml of %0,25 bupivacaine
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block
- Group P (Active Comparator): Participants who will be receiving a thoracal paravertebral block with a single dose of 30 ml of %0,25 bupivacaine
  Interventions: Procedure: Paravertebral Block

INTERVENTIONS:
Procedure: Serratus Posterior Superior Intercostal Plane Block — Before the induction of general anesthesia, under aseptic conditions, serratus posterior superior intercostal plane block will be performed with a single dose of 30 ml of %0,25 bupivacaine with ultrasound guidance, by the senior anaesthesiologist.
  Arms: Group S
Procedure: Paravertebral Block — Before the induction of general anesthesia, under aseptic conditions, paravertebral block will be performed with a single dose of 30 ml of %0,25 bupivacaine with ultrasound guidance, by the senior anaesthesiologist.
  Arms: Group P

SUMMARY:
The goal of this clinical trial is to compare the analgesic efficacy of thoracal paravertebral block (TPVB) and serratus posterior superior intercostal plane block (SPSIPB) in patients undergoing video-assisted thoracoscopic surgery (VATS). The main questions it aims to answer are:

How will the total perioperative opioid consumption of the patients receiving two different blocks change? How will TPVB and SPSIPB effect the patients' numeric rating scores for pain in the postoperative 24-hour period? How will TPVB and SPSIPB effect the incidence of opioid related side effects?

Participants will be divided in two groups:

TPVB group will receive a TPVB before the surgery. SPSIPB group will receive a SPSIPB nerve block before the surgery. Researchers will compare the results between the groups to see the postoperative effects concerning opioid consumption as well as the pain scores, respiratory parameters and opioid associated side effects.

The hypothesis of this study is that participants receiving SPSIPB for VATS will have a less total opioid consumption 24 hours postoperatively.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgeries require a surgical incision of the lateral thoracic wall. In order to ease the postoperative pain of patients undergoing VATS, some regional anaesthesia techniques have been tried but there is no consensus on the best method. The gold standard peripheric nerve block is considered to be thoracal paravertebral block (TPVB). Recently, a new nerve block called serratus posterior superior intercostal plane block (SPSIPB) has been described. The anatomic and radiologic studies of SPSIPB suggest that the local anaesthetic distributes from C7 to T10 vertebrates, covering the surgical site of VATS. This study aims to compare the analgesic efficacy of TPVB and SPSIPB for VATS. The hypothesis is that participants receiving SPSIPB for VATS will have a less total opioid consumption 24 hours postoperatively. Also, the postoperative pain scores and opioid related side effects of the participants will be recorded. Participants will be divided in two groups. The group P will receive a TPVB preoperatively in the operating room. The group S will receive a SPSIPB preoperatively in the operating room. The participants will be followed 24 hours postoperatively and their total opioid consumption, numeric rating scores for pain, incidence of opioid related side effects will be recorded. Also the participants and the surgical teams perioperative pain related satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-80 undergoing video-assisted thoracoscopic surgery

Exclusion Criteria:

* Allergy to local anaesthetics Chronic opioid use history Patients with psychiatric disorders Patients who are not open to communication Patients with chronic organ failure Patients that do not give consent Patients that need emergency surgery within the first 24 hours of the initial surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-03 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours post-surgery
  all consumed opioids will be converted in morphine equivalents and then added to reach the total dosage

SECONDARY OUTCOMES:
Numeric rating scale scores for pain | 24 hours post-surgery
  the scale between 0: no pain and 10:highes pain answered by the participants
Opioid related side effects | 24 hours post-surgery
  Nausea, vomiting, pruritis, respiratory depression assessed by yes/no questions

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Darçın, MD, Principal Investigator — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting from 6 months after publication for 5 years
Access Criteria: no access criteria